CLINICAL TRIAL: NCT03343210
Title: Quality of Life and Cancers in Nursing Homes
Acronym: QUALICE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: due to covid pandemic
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: QUALICE 16-180
Record Dates: First submitted 2017-03-07; First posted 2017-11-17 (Actual); Last update posted 2021-10-07 (Actual); Status verified 2020-01

CONDITIONS: Quality of Life; Cancer; Nurse's Role
MeSH Terms: conditions — Neoplasms | interventions — Pain Measurement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cancer patient (Experimental): cancer patient
  Interventions: Diagnostic Test: quality of life and pain measurement .
- no cancer patient (Active Comparator): no cancer patient
  Interventions: Diagnostic Test: quality of life and pain measurement .

INTERVENTIONS:
Diagnostic Test: quality of life and pain measurement . — comparison of quality of life measurement in residents with cancer and in cancer-free residents, by a geriatric consultations'nurse

SUMMARY:
Quality of life (QOL) of nursing homes residents with cancer in France is not known. High prevalence of neurodegenerative diseases makes it difficult. It was found that oncological management is suboptimal among Poitevin territory residents. Publications report an inadequate management of symptoms of discomfort related to cancers.

The multicentric study will comparate quality of life in patients with and without Cancers in nursing homes, including residents with neurodegenerative disease, using validated questionnaires. These questionnaires, as well as pain evaluation, will be carried out by a geriatric consultations' nurse.

DETAILED DESCRIPTION:
Investigators will also make a descriptive inventory of the oncological care and support care in these patients, in order to evaluate the need for a specific oncogeriatric intervention.

Quality of life and pain will be compared with a randomized residents control group, in each hospital.

ELIGIBILITY:
Inclusion Criteria:

* Affiliated to the social security system
* talking french language
* Cancer group: All residents with a history of cancer,
* Control group: residents without any history of cancer (same number of residents as in the cancer group), randomly selected in each nursing home, matched to age, sex, presence of dementia (mild or Moderate), and AGGIR dependancy scale

Exclusion Criteria:

* Severe dementia (MMS <10/30) • Total disability to communicate

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 73 (Actual)
Dates: Start 2018-07-18 (Actual); Primary Completion 2018-08-16 (Actual); Study Completion 2020-07-09 (Actual)

PRIMARY OUTCOMES:
quality of life measurement in patients | day 1
  Logsdon Quality Of Life Alzheimer Dementia scale if neurodegenerative disease or WHO-Quality Of Life- OLD scale if none

SECONDARY OUTCOMES:
pain level | day 1
  Simple Verbal Scale or Doloplus scale
independance loss | day 1
  AGGIR(Autonomie Gérontologique et Groupes Iso-Ressources) scale
frequency of dementia | 3 months
  in ordrer to Prepare a interventionnal care study for residents with cancer: Describing cancers management in nursing homes without any oncogeriatrician, Refining the expected effect of an oncogeriatry intervention on QOL (margin of improvement relative to the cancer free population) Estimating the intraclass correlation coefficient of QOL, Compare quality of life scores among seniors with no cognitive impairment

CONTACTS AND LOCATIONS:
Locations (6):
- France (6):
  - Amiens UH, Amiens
  - Caen UH, Caen
  - Pasteur HC, Cherbourg
  - Fecamp HC, Fécamp
  - Rouen UH, Rouen
  - Saint Quentin HC, Saint-Quentin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Drageset J, Corbett A, Selbaek G, Husebo BS. Cancer-related pain and symptoms among nursing home residents: a systematic review. J Pain Symptom Manage. 2014 Oct;48(4):699-710.e1. doi: 10.1016/j.jpainsymman.2013.12.238. Epub 2014 Apr 3. PMID 24703946
- [Result] Novella JL, Dhaussy G, Wolak A, Morrone I, Drame M, Blanchard F, Jolly D. [Quality of life in dementia: state of the knowledge]. Geriatr Psychol Neuropsychiatr Vieil. 2012 Dec;10(4):365-72. doi: 10.1684/pnv.2012.0375. French. PMID 23250016
- [Result] Leplege A, Perret-Guillaume C, Ecosse E, Hervy MP, Ankri J, von Steinbuchel N. [A new instrument to measure quality of life in older people: The French version of the WHOQOL-OLD]. Rev Med Interne. 2013 Feb;34(2):78-84. doi: 10.1016/j.revmed.2012.07.011. Epub 2012 Dec 23. French. PMID 23266010
- [Result] Wheelwright S, Darlington AS, Fitzsimmons D, Fayers P, Arraras JI, Bonnetain F, Brain E, Bredart A, Chie WC, Giesinger J, Hammerlid E, O'Connor SJ, Oerlemans S, Pallis A, Reed M, Singhal N, Vassiliou V, Young T, Johnson C. International validation of the EORTC QLQ-ELD14 questionnaire for assessment of health-related quality of life elderly patients with cancer. Br J Cancer. 2013 Aug 20;109(4):852-8. doi: 10.1038/bjc.2013.407. Epub 2013 Jul 18. PMID 23868003